CLINICAL TRIAL: NCT05377801
Title: Multifaceted Fall Prevention Program for Chinese Community-dwelling Older Adults With Fall Risks: A Pilot Randomized Controlled Trial
Brief Title: Chinese Version of LIVE-LiFE for Older Adults With Previous Falls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sigma Theta Tau International (Other)
Responsible Party: Principal Investigator, Minhui Liu, Associate professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00186421
Record Dates: First submitted 2021-12-16; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Accidental Falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group of this study is a multi-dimensional intervention conducted by nursing students over a 12-week period, consisting of four parts: individualized balance and strength training, vision screening, drug evaluation, home risk assessment and home repair and transformation. These components were carried out through a combination of personal home visits and telephone interviews.
  Interventions: Behavioral: Multi-dimensional fall prevention intervention program for 12 weeks
- The control group (No Intervention): The control group would receive the same amount of health education.

INTERVENTIONS:
Behavioral: Multi-dimensional fall prevention intervention program for 12 weeks — The intervention group of this study is a multi-dimensional intervention conducted by nursing students over a 12-week period, consisting of four parts: individualized balance and strength training, vision screening, drug evaluation, home risk assessment and home repair and transformation. These components were carried out through a combination of personal home visits and telephone interviews.
  Arms: The intervention group

SUMMARY:
The research is to solve the problem of the high incidence of falls among older adults in China. To this end, the investigators will develop a multi-dimensional fall prevention program by cultivating nursing students as community intervention personnel to address the current shortage of fall prevention programs and professional intervention in China. The research will make an important contribution to health care.

DETAILED DESCRIPTION:
The study intervention group is a 12-week multi-dimensional intervention, consisting of four parts: individualized balance and strength training, vision screening, drug evaluation, home risk assessment and home repair and transformation. Interventors will teach skills related to balance and strength training, incorporate these principles and exercises into daily and leisure activities, and how to increase the challenge of balance. The one-hour home visit aims to develop a personalized plan for participants by understanding each participant's health, exercise preferences, sedentary behaviors, and identifying needs related to the risk of falling. In particular, the interventionist will work with the participant to determine 6 skills or activities, and the participant hopes to practice ankle weight bearing at least 3 times a week based on their interests and abilities. Interventions and participants will work together to develop personal goals and plans, using exercise logs for gradual exercise, to continuously increase strength, resistance, weight, and challenge balance or strength. During home visits, the intervener will also assess participants' inherent risks by assessing their visual acuity, assess their home risk factors, and discuss with their caregiver or their children what risks would arise if the elderly live alone. In addition to group meetings and home visits, the interventionists will call to ask about progress and provide support and encouragement. Participants in the control group will receive the same amount of health education。

ELIGIBILITY:
Inclusion criteria:

* age ≥60 years;
* Falls ≥2 times or injuries caused by falls ≥ 1times in the past year;

Exclusion criteria:

* residents who cannot live in a community in Changsha for more than 3 months, or who reside in a long-term care institution in Changsha;
* Moderate to severe cognitive impairment based on a simple and portable mental state questionnaire;
* Unable to walk independently;
* Has the nervous system condition which seriously affects its gait and activity;
* Any unstable or terminal illness that may interfere with planned exercise and is unlikely to be resolved;
* He is currently undergoing physical therapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Physical Functioning:1.（short physical performance battery, SPPB） | Three months
  SPPB is used to evaluate the comprehensive functions of lower limb muscle strength, balance, and walking, including 3 parts: 5 sit-ups, standing in series (including two feet standing side by side, one heel and the other side of the big toe standing sideways, one Stand with the heel of one foot close to the top of the big toe of the other foot) and walk 8 feet.
Physical Functioning:2. (timed get up and go test/the timed up and go test, TUG) | Three months
  2. TUG involves balance in the sitting position, whether the transition from sitting to standing is smooth, walking gait, speed, and stability, and whether hesitant to turn around, etc., and can be used to evaluate the dynamic balance ability and mobility function.

SECONDARY OUTCOMES:
Fear of falling was assessed by the Fall Efficacy Scale-International Chinese Version (FES-I (Ch)) Fear of falls was assessed by the Fall Efficacy Scale-International Chinese Version (FES-I (Ch)) | Three months
  FES-I (Ch) measures the degree of anxiety about falls among participants during 16 activities. The total score ranges from 16-64 points, a higher total score indicates a greater sense of fall efficacy. The original FES-I and FES-I (Ch) have good reliability (Cronbach's alpha: 0.96 ~ 0.97) and have structural validity in different studies.
Quality of life was measured using the Chinese version of the five EuroQol questionnaire (EQ-5D) | Three months
  Participants will be asked if they have no problems in five dimensions, some or moderate questions, including actions, self-care, daily activities, pain / discomfort, anxiety / depression. The total score ranges from 0 to 100 points, higher scores mean a better quality of life.
Cognitive function and mental status are adopted: Mini-cog Test, Patient health questionnaire (PHQ-9). | Three months
  (1) Mini-cog Test, which can be completed in 3 minutes, and is mostly used to distinguish whether or not they have dementia. The total score ranges 1 to 3, higher scores mean a better cognitive status. The scale has a sensitivity of 76% ～ 99%, specificity is 89% -93%, and has a good predictive value of dementia for the participants. (2) Patient health questionnaire (PHQ-9). This scale is used to understand how much time participants have been affected by 9 questions including depression and interest in the past two weeks. The total score ranges from 0 to 27, higher scores mean a worse depressive status. The researchers Summarized (PHQ-9) that the Cronbach's alpha used in the community elderly population was 0.832, the sensitivity was 88%, and the specificity was 99% 49.
Living habits and physical activities used: Physical Activity Scale for the Elderly (PASE), Activity of daily living function (ADL), Instrumental Daily Life Activity Ability Scale (IADL) | Three months
  (1) Physical Activity Scale for the Elderly (PASE). The scale consists of 10 major categories of problems, including physical exercise, housework, and occupational physical activity. The total score range from 0 to 400, higher scores mean a better physical activity. (2) Activity of daily living function (ADL), which includes two parts: Physical Self-Maintenance Scale (PSMS; 6 items) and instrumental ability of daily living Scale (Instrumental Activity of Daily Living IADL; 8). Each entry is graded on a scale of 1 to 4. The total score ranges from 0 to 100, higher scores mean a worse ability of daily activity. (3) Instrumental Daily Life Activity Ability Scale (IADL): Includes recreation and leisure, use of transportation, cooking, housework maintenance, telephone use, medication, and financial management. The total score ranges from 0 to 56, higher scores mean a worse ability of instrumental daily activity.
Taking medications and dietary supplements uses the Beliefs About Medical Questionnaire (BMQ) | Three months
  Medical Questionnaire (BMQ), which includes two sub-scales: the patient's general belief in any drug (BMQ-General) and specificity for a certain class of drugs Belief (BMQ-Specific). The researchers experimentally obtained the Cronbach's alpha coefficients of the two dimensions of the Chinese version of BMQ medication necessity and medication concern in elderly patients with depression; the retest reliability was 0.743 and 0.786, respectively; Degree coefficient (CVI) is 0.80 ~ 1.00

CONTACTS AND LOCATIONS:
Overall Officials: Minhui Liu, Ph.D, Principal Investigator — Central South University
Locations (1):
- Central South University, Changsha, Hunan, China